CLINICAL TRIAL: NCT02433496
Title: Physician Coaching to Reduce Opioid-related Harms
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Center for Health Enhancement System Studies (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0280; 1R34DA036720-01A1 (NIH)
Record Dates: First submitted 2015-04-20; First posted 2015-05-05 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Substance Abuse; Chronic Pain
Keywords: Opioid
MeSH Terms: conditions — Substance-Related Disorders; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Physician coaching: This group includes 4 intervention primary care clinics that are part of the University of Wisconsin's Department of Family Medicine. These clinics will receive an organizational coaching intervention that includes in-person site visits and phone/email communication. Each participating clinic will designate one primary care physician to act as a clinic lead in working with the coach to coordinate an initial site visit (during project month 13, July 2015), a follow-up site visit (month 15, October, 2015), and communicating with the coach throughout the 6-month follow-up period via phone and email.
  Interventions: Other: Physician coaching
- Control Group: This group includes 4 control primary care clinics that will not receive any intervention. A de-identified dataset will be created to examine differences in outcome variables between intervention and control clinics.

INTERVENTIONS:
Other: Physician coaching — The coach will present the latest research on the benefits and risks of long-term opioid use. The presentation will be followed by a brainstorming exercise where the coach joins the clinic team in experiencing clinical practices from the perspective of a patient with chronic pain. The coach will help the clinic team flowchart clinical workflows and determine the best course for implementing aspects of a checklist-based implementation guide developed to support adoption of the guidelines for opioid prescribing.
  The coach will help the team implement ideas using Plan-Do-Study-Act change cycles. The coach will maintain monthly email and phone contact with the clinic lead and clinic team after the initial site visit to monitor implementation progress and offer advice.
  Groups: Physician coaching

SUMMARY:
This project pilot tests an innovative clinical guideline translation and physician coaching model to promote adherence to evidence-based guidelines for the prescribing of opioid pain medications in primary care settings.

DETAILED DESCRIPTION:
This project addresses the urgent need to promote the adoption of evidence-based practices in healthcare by pilot-testing an innovative implementation strategy. The implementation strategy aims primarily to reduce variation in opioid prescribing practices for chronic pain in primary care settings.

The standard approach to improving medical practice involves groups of clinical experts reviewing the literature to produce clinical guidelines based on scientific evidence, and disseminating those guidelines by publishing them in medical journals. A clinical guideline has been developed for opioid prescribing for chronic non-cancer pain using this type of approach. The implementation strategy for promoting uptake of the guideline in primary care settings tested in this study consists of three innovations: (1) a process for translating clinical guidelines into a checklist-based implementation guide for clinicians, (2) a physician peer coaching model, and (3) implementation support using tools from systems engineering. This project teams the experts who developed the guideline for opioid prescribing with experts in implementation science and primary care to translate the guideline into an actionable, checklist-based implementation guide. If the implementation strategy is effective in this pilot test, it will be used in a larger cluster-randomized trial to test it against other approaches to evidence-based practice adoption.The long-term goal of this research is to improve the adoption of evidence-based practices in primary care by producing a generalizable model of change.

ELIGIBILITY:
Inclusion Criteria:

At each of the 4 coaching intervention sites, we aim to recruit between 3-7 clinical care providers with prescribing authority (e.g., primary care physicians, mid-level practitioners, etc.) to participate in interviews and focus groups. All clinic staff (e.g., medical assistants, office staff) are welcome to participate in coaching site visits and follow up correspondence, but only staff with prescribing authority will be considered research participants.

Exclusion Criteria:

* Residents will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinicians with prescribing authority at community-based primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 53132 (Actual)
Dates: Start 2014-07; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R Quanbeck, PhD, Principal Investigator — Center for Health Enhancement Systems Studies
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Quanbeck A, Brown RT, Zgierska AE, Jacobson N, Robinson JM, Johnson RA, Deyo BM, Madden L, Tuan WJ, Alagoz E. A randomized matched-pairs study of feasibility, acceptability, and effectiveness of systems consultation: a novel implementation strategy for adopting clinical guidelines for Opioid prescribing in primary care. Implement Sci. 2018 Jan 25;13(1):21. doi: 10.1186/s13012-018-0713-1. PMID 29370813

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Clinics were paired and randomly assigned to be grouped in the intervention or control group. The intervention group was invited. If clinics in this group refused to participate, the other clinic of the pair was invited to be a part of the intervention group. Once clinics agreed to take part in the study they were immediately assigned to a group.
Units Other Than Participants: clinics
Groups:
- Physician Coaching: This group included 4 intervention primary care clinics that received an organizational coaching intervention that included in-person site visits and phone/email communication. Each participating clinic was designated one primary care physician to act as a clinic lead in working with the coach to coordinate an initial site visit, a follow-up site visit, and communicating with the coach throughout the 6-month follow-up period.
  Physician coaching: The coach presented the latest research on the benefits and risks of long-term opioid use. The coach helped the clinic team flowchart clinical workflows and determined the best course for implementing aspects of a checklist-based implementation guide developed to support adoption of the guidelines for opioid prescribing.
  The coach helped the team implement ideas using Plan-Do-Study-Act change cycles and maintained contact with the clinic lead and clinic team after the initial site visit to monitor implementation progress and offer advice.
- Control Group: This group included 4 control primary care clinics that did not receive any intervention. A de-identified dataset was created to examine differences in outcome variables between intervention and control clinics.
- Refused Group: Clinics were invited to join the study, but refused to receive the intervention. Clinics reason for refusal was lack of staff or time. Data was not collected or analyzed for clinics that refused the intervention.
Period: Overall Study
Arm/Group | Physician Coaching | Control Group | Refused Group
Started | 29990; 4 clinics (This includes patients (29956) and providers (34).) | 13309; 4 clinics (This includes patients (13296) and providers (13).) | 9833; 3 clinics (This includes patients (9813) and providers (20).)
Completed | 29990; 4 clinics (This includes patients (29956) and providers (34).) | 13309; 4 clinics (This includes patients (13296) and providers (13).) | 9833; 3 clinics (This includes patients (9813) and providers (20).)
Not Completed | 0; 0 clinics | 0; 0 clinics | 0; 0 clinics

BASELINE CHARACTERISTICS:
Population: Participants include patients and providers. Patient counts for Physician coaching, Control Group, and Refused group were 29956, 13296, and 9813, respectively. Provider counts for Physician coaching, Control Group, and Refused group were 34, 13, and 20, respectively.
Units Other Than Participants: clinics
Groups:
- Refused Group: This group included 3 primary care clinics that were approached to participate in the study, but refused to participate.
- Total: Total of all reporting groups
Arm/Group | Physician Coaching | Control Group | Refused Group | Total
Number analyzed (Participants) | 29990 | 13309 | 9833 | 53132
Number analyzed (clinics) | 4 | 4 | 3 | 11
Age, Customized [Count of Participants; unit: Participants]
  Age of participants: < 18 years old | 0 | 0 | 0 | 0
  Age of participants: >= 18 years old | 29990 | 13309 | 9833 | 53132
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14125 | 6615 | 4504 | 25244
  Male | 15865 | 6694 | 5329 | 27888
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 660 | 333 | 246 | 1239
  Not Hispanic or Latino | 29330 | 12976 | 9587 | 51893
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 150 | 67 | 49 | 266
  Asian | 720 | 213 | 69 | 1002
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 720 | 306 | 69 | 1095
  White | 24831 | 11126 | 8525 | 44482
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3569 | 1597 | 1121 | 6287
Proportion of patients with consistent opioid Rx [Number; unit: proportion of patients] — Population: This measure analyzes at the patient level. The population not analyzed for this measure are providers of the clinic. The Refused group was not analyzed due to desire not to participate in the study.
  proportion of patients
    number analyzed (Participants) | 29956 | 13296 | 0 | 43252
    (all) | 0.013 | 0.014 |  | 0.013
Proportion with mental health screen [Number; unit: proportion of patients] — Population: This measure analyzes at the patient level and includes only the subset of patients with consistent opioid Rx.
  proportion of patients
    number analyzed (Participants) | 389 | 186 | 0 | 575
    (all) | 0.226 | 0.220 |  | 0.224
Proportion with urine drug screen [Number; unit: proportion of patients] — Population: This measure analyzes at the patient level and includes only the subset of patients with consistent opioid Rx.
  proportion of patients
    number analyzed (Participants) | 389 | 186 | 0 | 575
    (all) | 0.399 | 0.374 |  | 0.391
Proportion with treatment agreement [Number; unit: proportion of patients] — Population: This measure analyzes at the patient level and includes only the subset of patients with consistent opioid Rx.
  proportion of patients
    number analyzed (Participants) | 389 | 186 | 0 | 575
    (all) | 0.428 | 0.368 |  | 0.409
Average morphine equivalent daily dose (MEDD) [Mean (Standard Deviation); unit: milligram] — Population: This measure analyzes at the patient level and includes only the subset of patients with consistent opioid Rx.
  milligram
    number analyzed (Participants) | 389 | 186 | 0 | 575
    (all) | 86.3 (18.7) | 58.8 (10.1) |  | 72.5 (16.9)
Proportion with MEDD >120 mg [Number; unit: proportion of patients] — Population: This measure analyzes at the patient level and includes only the subset of patients with consistent opioid Rx.
  proportion of patients
    number analyzed (Participants) | 389 | 186 | 0 | 575
    (all) | 0.215 | 0.137 |  | 0.190
Proportion with co-prescribed benzodiazepines [Number; unit: proportion of patients] — Population: This measure analyzes at the patient level and includes only the subset of patients with consistent opioid Rx.
  proportion of patients
    number analyzed (Participants) | 389 | 186 | 0 | 575
    (all) | 0.08 | 0.055 |  | 0.072

OUTCOME MEASURES:

1. Primary Outcome: Overall Rate of Opioid Prescribing
Description: The proportion of patients with a chronic pain diagnosis receiving daily opioids.
Time Frame: Up to 3 years
Population: This is the number of patients in each group.
Measure: Number; unit: Proportion of patients
Arm/Group | Physician Coaching | Control Group
Number analyzed (Participants) | 29956 | 13296
Proportion of patients | 0.012 | 0.013

2. Secondary Outcome: Rate of Opioid / Benzodiazepine Co-prescribing
Description: Proportion of patients with a chronic pain diagnosis receiving daily opioids and benzodiazepines concurrently.
Time Frame: Up to 3 years
Population: This is the number of patients who fall in the subset of consistent opioid use.
Measure: Number; unit: Proportion of patients
Arm/Group | Physician Coaching | Control Group
Number analyzed (Participants) | 359 | 160
Proportion of patients | 0.074 | 0.061

3. Secondary Outcome: Urine Drug Screening Rate
Description: Proportion of opioid patients completing urine drug screens prior to and during the study intervention
Time Frame: Up to 3 years
Population: This is the number of patients who fall in the subset of consistent opioid use.
Measure: Number; unit: Proportion of patients
Arm/Group | Physician Coaching | Control Group
Number analyzed (Participants) | 359 | 160
Proportion of patients | 0.645 | 0.440

4. Secondary Outcome: Mental Health Screening Rate
Description: Proportion of opioid patients screened for mental health/substance use problems
Time Frame: Up to 3 years
Population: This is the number of patients who fall in the subset of consistent opioid use.
Measure: Number; unit: Proportion of patients
Arm/Group | Physician Coaching | Control Group
Number analyzed (Participants) | 359 | 160
Proportion of patients | 0.574 | 0.394

5. Secondary Outcome: Use of Pain Management Agreements
Description: Proportion of opioid patients signing pain management agreements
Time Frame: Up to 3 years
Population: This is the number of patients who fall in the subset of consistent opioid use.
Measure: Number; unit: Proportion of patients
Arm/Group | Physician Coaching | Control Group
Number analyzed (Participants) | 359 | 160
Proportion of patients | 0.782 | 0.542

6. Secondary Outcome: High-dose Patients
Description: Proportion of opioid prescriptions above 120 mg daily morphine equivalent
Time Frame: Up to 3 years
Population: This is the number of patients who fall in the subset of consistent opioid use.
Measure: Number; unit: Proportion of patients
Arm/Group | Physician Coaching | Control Group
Number analyzed (Participants) | 359 | 160
Proportion of patients | 0.191 | 0.125

7. Secondary Outcome: Provider Drop-out Rate
Description: Number and percentage of providers who drop out of study at 3 months
Time Frame: 3 months
Population: This is at the prescriber level.
Measure: Count of Participants; unit: Participants
Arm/Group | Physician Coaching | Control Group
Number analyzed (Participants) | 34 | 13
Participants | 0 | 0

8. Secondary Outcome: Participating Patient Demographics
Description: Characteristics of participating patients vs. general patient population (race, gender, ethnicity)
Time Frame: Up to 3 years
Measure: Number; unit: percentage of patients
Arm/Group | Physician Coaching | Control Group
Number analyzed (Participants) | 29956 | 13296
percentage of patients
  % female | 47.1 | 49.7
  % hispanic | 2.2 | 2.5
  % asian | 2.4 | 1.6
  % black | 2.4 | 2.3
  % native | 0.5 | 0.5
  % other | 11.9 | 12.2
  % white | 82.8 | 83.6

9. Secondary Outcome: Participating Clinic Characteristics
Description: Characteristics of participating clinics vs. non-participating clinics (number of patients, number of providers, overall opioid prescribing rate)
Time Frame: Up to 12 months
Measure: Number; unit: participants
Arm/Group | Physician Coaching | Control Group | Refused Group
Number analyzed (Participants) | 29990 | 13309 | 9833
participants
  number of patients | 29956 | 13296 | 9813
  number of providers | 34 | 13 | 20
  overall opioid prescribing rate | 359 | 160 | NA — Refused clinic data could not be obtained and analyzed.

10. Secondary Outcome: Participating Staff Characteristics
Description: Characteristics of participating staff (profession)
Time Frame: Up to 12 months
Population: These are clinic staff that made up the clinic change teams. Since change teams were specific to the physician coaching group, no change teams were constructed in the Control group, thus there is no data to be reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Physician Coaching
Number analyzed (Participants) | 27
Participants
  Medical doctor | 6
  Nurse practitioner | 1
  Registered nurse | 4
  Licensed practical nurse | 3
  Clinic operations assistant | 1
  Clinic operations manager | 2
  Lab staff | 2
  Reception | 3
  Medical assistant | 5

11. Secondary Outcome: Intervention Fidelity
Description: Total hours of coaching delivered/received among all clinics that received physician coaching.
Time Frame: Up to 12 months
Population: Four clinics were analyzed for this measure. Since the intervention was specific to the physician coaching group, no time was spent in the Control group, thus there is no data to be reported.
Measure: Number; unit: hours spent delivering implementation
Units Other Than Participants: clinics
Arm/Group | Physician Coaching
Number analyzed (Participants) | NA
Number analyzed (clinics) | 4
hours spent delivering implementation
  Facilitator hours | 237.7
  physician consultant hours | 85.7

12. Secondary Outcome: Intervention Cost
Description: Total cost of coaching intervention among all clinics that received physician coaching. At clinic level.
Time Frame: Up to 12 months
Population: Four clinics were analyzed. No intervention was given to control group clinics, so there is no reported data.
Measure: Number; unit: Dollars
Units Other Than Participants: clinics
Arm/Group | Physician Coaching
Number analyzed (Participants) | NA
Number analyzed (clinics) | 4
Dollars | 29379

13. Secondary Outcome: Proportion With MEDD >120 mg
Description: The proportion of patients who have consistent opioid Rx above a morphine equivalent daily dose about 120 mg.
Time Frame: Up to 12 months
Population: This is the number of patients who have a consistent opioid Rx.
Measure: Number; unit: Proportion of participants
Arm/Group | Physician Coaching | Control Group
Number analyzed (Participants) | 389 | 186
Proportion of participants | 0.191 | 0.125

14. Secondary Outcome: Average Morphine Equivalent Daily Dose (MEDD)
Description: The average MEDD in milligrams for patients with consistent opioid Rx.
Time Frame: Up to 12 months
Population: This is the number of patients who have a consistent opioid Rx.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Physician Coaching | Control Group
Number analyzed (Participants) | 389 | 186
milligrams | 84.3 (16.8) | 60.2 (20.1)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the span of the study, 3 years.
Description: Because the intervention of this study was aimed at changing prescribing practices of providers, adverse events of patients treated at the clinics were not collected. Only adverse events of providers were collected.
Arm/Group | Physician Coaching | Control Group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/13
Other Adverse Events (participants affected / at risk) | 0/34 | 0/13

LIMITATIONS AND CAVEATS:
The UWHealth system introduced a new opioid-prescribing policy concurrent with the beginning of the study period and included a standardized treatment agreement that included elements of the checklist developed during this research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT02433496/Prot_SAP_000.pdf